CLINICAL TRIAL: NCT06245434
Title: Circadian Rhythmicity During Coma Awakening
Acronym: COMARHYTHM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL23_0053
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Acute Brain Injury Coma
Keywords: Circadian rhythms; Consciousness; Wakefulness; Biomarkers; Monoamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Main group with acute brain injury and initial Disorders of consciousness (Experimental): 50 patients in the initial phase of acute brain injury with disturbed consciousness, hospitalized in the Neurological Intensive Care Unit and at risk of delayed awakening
  Interventions: Behavioral: Repeated behavioural assessment; Behavioral: Act-Pass paradigm; Behavioral: Biological measures of circadian and monoamines biomarkers; Behavioral: Transcriptomic and genomic analysis; Behavioral: Polysomnography with concomitant environment recording; Behavioral: Actimetry; Behavioral: Morphological MRI; Behavioral: Assessment of correlation between patients' behaviour and neurophysiological markers of consciousness.
- Comparative group with acute brain injury without Disorders of consciousness (Active Comparator): 20 patients in the initial phase of brain damage WITHOUT disturbance of consciousness, hospitalized in the Neurological Intensive Care Unit and presenting similar causes of brain damage.
  Interventions: Behavioral: Repeated behavioural assessment; Behavioral: Act-Pass paradigm; Behavioral: Biological measures of circadian and monoamines biomarkers; Behavioral: Transcriptomic and genomic analysis; Behavioral: Polysomnography with concomitant environment recording; Behavioral: Actimetry; Behavioral: Morphological MRI; Behavioral: Assessment of correlation between patients' behaviour and neurophysiological markers of consciousness.
- Comparative group with post-acute Disorders of consciousness (Active Comparator): 20 patients in the sub-acute or chronic phase of a consciousness disorder and admitted to the Post-Resuscitation Rehabilitation Service.
  Interventions: Behavioral: Repeated behavioural assessment; Behavioral: Act-Pass paradigm; Behavioral: Biological measures of circadian and monoamines biomarkers; Behavioral: Transcriptomic and genomic analysis; Behavioral: Polysomnography with concomitant environment recording; Behavioral: Actimetry; Behavioral: Morphological MRI; Behavioral: Assessment of correlation between patients' behaviour and neurophysiological markers of consciousness.

INTERVENTIONS:
Behavioral: Repeated behavioural assessment — One CRS-R per visit
  * 4 SECONDs
  * Eye tracking during every clinical assessment
  * Recording every 2-4h of the Glasgow Coma Score
  * Recording every 2h of the temperature and pupillometer reactivity to light
Behavioral: Act-Pass paradigm — Before and after sedation withdrawal Assessment of infra-clinical response to an active paradigm (attention focalisation or diversion).
Behavioral: Biological measures of circadian and monoamines biomarkers — Systematic urinary sampling every 2 hours for melatonin, cortisol and monoamines metabolites
Behavioral: Transcriptomic and genomic analysis — Definition of the peripheral cellular clock by 2 transcriptomic measures Constitution of a genomic biobank to analyse the cofounding factors for circadian disruption and differential clinical recovery
Behavioral: Polysomnography with concomitant environment recording — One 48h polysomnography for the first visit
  + 3* 24h polysomnography for each visit Synchronised recordings of light, sound, activity in patients' rooms
Behavioral: Actimetry — Continuous recording of movements at the wrist during 7 days after sedation withdrawal
Behavioral: Morphological MRI — Precise description of brain lesion by a 3T MRI within the 1st week after sedation withdrawal
Behavioral: Assessment of correlation between patients' behaviour and neurophysiological markers of consciousness. — Video recording of spontaneous patients' movements in the bed and synchronized during 2h with high-density EEG.

SUMMARY:
Acute brain injury is a major cause of admission to intensive care units, as well as of mortality and morbidity, worldwide and for all age groups. With most patients surviving these injuries thanks to recent medical advances, society is facing not only the growing burden of disability, but above all the ethical issues involved in withdrawal of life-sustaining therapies (WSLT). To resolve this dilemma, effective treatment would be necessary, but this is hampered by our limited knowledge of the pathophysiological mechanisms of the natural history of coma, from onset to recovery. A more systematic description of coma awakening using a multimodal battery in intensive care unit patients would enable us to refine the awakening and re-emergence of consciousness and define appropriate biomarkers for selecting candidates in interventional studies.

The investigators hypothesize that the current postulate of successive stages (i.e. from one clinical class to the next) of coma recovery is incomplete, as it does not take into account the rhythmic nature of wakefulness. The investigators propose that the best correlate of the natural history of coma recovery is a gradual shift from the loss of physiological cycles to a circadian rhythmicity of arousal indices (behavioural and neurophysiological) and a wide amplitude of metric fluctuations in assessing content richness.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Admission to the Neurological Intensive Care Unit
* Initial disorder of consciousness (GCS < 8) or initial brain lesion (on CT or MRI) requiring intubation and sedation during management (for upper airway protection or due to coma)
* Intubated patient under mechanical ventilation wwith no response to simple commands
* Weaning from sedation : acquired / possible within 7 days of inclusion in the absence of new complications
* Severity of clinical or morphological impairment leading to risk of persistent disturbance of consciousness
* Sedation discontinued or able to be discontinued within 3 month of initial management of the disorder of consciousness or brain injury
* Effective treatment of the cause of admission without risk of short-term recurrence
* Patient aged 17 or over
* Urinary catheter in place at the time of inclusion and to remain in place until Visit N°1
* Presence of relatives able to sign consent or of the minor's legal representative

Group 2

* Admission to the Neurological Intensive Care Unit or the Neurological Continuing Care Unit
* Absence of severe disorder of consciousness but possibility of minimal alteration of the initial Glasgow score (GCS between 9 and 15) with no time limit, with a stratification of three consecutive patient populations distinguished by the initial neurological alteration:

  * GCS = 15
  * GCS < 15 by predominance of an initial defect in responses to simple or complex commands obtained by motor or verbal means, without abnormality of arousal (E score = 4 but M score < 6 and/or V score < 5)
  * GCS < 15 with predominant initial somnolence, with or without abnormal motor or verbal responses to simple or complex commands (E score = 2 or 3 but M score = 6 and/or V score = 5).
* Existence of functional communication or functional use of objects at inclusion
* Mechanism of injury for which the aetiology is no longer active or at risk of recurrence
* Patient aged 17 or over
* Urinary catheter in place at the time of inclusion and to remain in place until Visit N°1
* In the case of impaired judgement despite functional communication or in the case of aphasia with functional use of objects: presence of relatives able to sign consent or of the legal representative of the minor or of the legal representative of the protected adult.

Group 3

* Admission to the Adult Post-Resuscitation Rehabilitation Department, in the Neurological Multidisciplinary Intensive Care Unit
* Disturbance of consciousness defined by an absence of communication or an absence of functional use of objects (for patients with aphasia), i.e. the two signs that could indicate emergence from the pauci-relational state, which includes patients presenting :

  * persistent coma
  * a vegetative state (or unresponsive wakefulness syndrome)
  * a pauci-relational state (MCS- or MCS+ if responding to simple commands).
* Persistent within the following timeframe

  * More than 3 months after the initial management of the disorder of consciousness or brain injury
  * More than 1 month after a post-anoxic coma.
* Mechanism of injury for which the aetiology is no longer active or at risk of recurrence
* Patient aged 17 or over
* Presence of relatives likely to sign the consent or of the legal representative of a minor or of the legal representative of a protected adult

Exclusion Criteria:

Group 1

* Subjects with a contraindication to MRI scans
* Admission for status epilepticus
* Existence of status epilepticus during the stay and persisting for > 24h or presenting an electrical remission for less than 48h prior to inclusion
* Post-anoxic coma with bilateral abolition of N20 PES cortical responses
* Coma related to a potentially recurrent cause of coma (tumours, infectious diseases with risk of relapse and inflammatory diseases)
* Moribund patient (life expectancy < 24h) or in WLST (no assessment possible of the dynamics of ongoing awakening)
* Haemodynamic or respiratory instability incompatible with a prolonged attempt to stop sedation (except in the case of scheduled surgery outside the visit dates)
* Patients under guardianship, curatorship or safeguard of justice
* Patients not affiliated to the French health insurance system
* Pregnant women or women of childbearing age without proof of the absence of a current pregnancy

Group 2

* Subjects with a contraindication to MRI scans
* Epileptic seizures on admission or during the stay

  * Single seizure: if no rapid return to consciousness (GCS < 8 for > 12 hours)
  * > 2 distinct epileptic seizures regardless of the duration of loss of consciousness
  * Status epilepticus
* Post-anoxic coma with bilateral abolition of N20 cortical PES responses.
* Coma linked to a potentially recurrent cause of coma (tumour, infection with risk of relapse and inflammation).
* A moribund patient (life expectancy < 24 hours) or a patient undergoing WLST with a high risk of death before the end of the study (inclusion possible if no therapeutic escalation is decided in a stabilised patient).
* Haemodynamic or respiratory instability incompatible with prolonged evaluation of the absence of sedation (risk of general anaesthesia for further failure, except in the case of scheduled surgery outside the visit dates).
* Patients under guardianship, curatorship or safeguard of justice
* Patients not affiliated to the French health insurance system
* Pregnant women or women of childbearing age without proof of the absence of a current pregnancy

Group 3

* Subjects with a contraindication to MRI scans
* Epileptic seizures during the week preceding inclusion:

  * Single seizure: if no rapid return to usual state of consciousness for > 12 hours
  * > 2 separate comitial seizures regardless of duration of loss of consciousness
  * Epileptic malaise
* Post-anoxic coma with bilateral abolition of N20 cortical responses to SEP
* Coma related to a potentially recurrent cause of coma (tumour, infection with risk of relapse and inflammation)
* Moribund patients (life expectancy < 24 hours) or patients undergoing WSLT with a high risk of death before the end of the study (inclusion possible if no therapeutic escalation is decided in a stabilised patient).
* Haemodynamic or respiratory instability incompatible with prolonged evaluation of the absence of sedation (risk of general anaesthesia for further failure, except in the case of scheduled surgery outside the visit dates).
* Patients under guardianship, curatorship or safeguard of justice prior to the event that provoked their state of chronic disturbance of consciousness. Patients under guardianship because of their chronic disorder of consciousness are eligible for the study.
* Patients not affiliated to the French health insurance system
* Pregnant women or women of childbearing age without proof of the absence of a current pregnancy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2028-12-02 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Consciousness outcome | 2, 3, 4,6 months post injury
  Coma Recovery Scale - revised used to define 4 possible consciousness outcomes (the best observed before death if the patient died at the date of assessment):
  * Coma
  * Unresponsive Wakefulness Syndrome
  * Minimally Conscious State
  * Exit-Minimally Conscious State (conscious patient)

SECONDARY OUTCOMES:
Functional outcome | GOS: 2, 3, 4,6 months post injury GOSE: 6 months post injury
  Glasgow Outcome Scale (GOS) Glasgow Outcome Scale Extended (GOSE)
  Minimum score 1 and maximum score 5. The lowest score is 5.
Cognitive outcome | 6 months post injury
  MOCA scale
  The MOCA is a short 30-question test that assesses several cognitive domains and allows for early detection of cognitive disorders. The MOCA test takes about 10-15 minutes to administer and consists of several sections, the first of which is an assessment of orientation in time and space. Then there are tasks that assess memory, concentration and reasoning ability, as well as language and visuospatial ability tasks.
  The MOCA score can range from 0 to 30 points, with a score of 26 points or more considered normal.
Quality of life outcome SF-36 scale | 6 months post injury
  At the end, a score for each dimension of the SF-36 was calculated, ranging from 0 to 100. A low score reflects a perception of poor health, loss of function, presence of pain. A high score reflects a perception of good health, absence of functional deficit, and pain (3,6,7)

CONTACTS AND LOCATIONS:
Overall Officials: GOBERT FLORENT, M.D. Ph.D., Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de Réanimation Polyvalente Neurologique Hôpital Neurologique Pierre Wertheimer, Bron, Lyon, France